CLINICAL TRIAL: NCT06052527
Title: Autonomous Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) and Influenza Treatment System With Machine Learning in Outpatient Settings
Brief Title: Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) and Influenza Treatment System With Machine Learning
Status: Completed | Type: Observational
Sponsor: Lizora LLC (Industry)
Collaborators: Sheng'ai Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Liz2023Covid19
Record Dates: First submitted 2023-09-21; First posted 2023-09-25 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; Post-COVID-19 Syndrome; Influenza
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active Covid-19 Infection: Patients with positive SARS-CoV-2 rapid antigen test results within 60 days before the start of the study will be administered pre-defined TCM prescriptions recommended by the Autonomous Treatment System based on machine learning
  Interventions: Other: Autonomous Treatment System for Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection and Influenza Based on Machine Learning
- Post-Covid-19 Syndrome: Patients with positive Covid-19 antigen test results obtained more than 60 days before the start of the study will be administered pre-defined TCM prescriptions recommended by the Autonomous Treatment System based on machine learning.
  Interventions: Other: Autonomous Treatment System for Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection and Influenza Based on Machine Learning
- Influenza: Patients with negative SARS-CoV-2 rapid antigen test results and who are diagnosed with influenza will be administered pre-defined TCM prescriptions recommended by the Autonomous Treatment System based on machine learning.
  Interventions: Other: Autonomous Treatment System for Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection and Influenza Based on Machine Learning

INTERVENTIONS:
Other: Autonomous Treatment System for Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection and Influenza Based on Machine Learning — A novel treatment recommendation system for Covid-19, Post-Acute Sequelae of SARS-CoV-2 Infection and Influenza, which is based on machine learning

SUMMARY:
This is an open-tabled, one-arm observatory trial to assess the effectiveness and safety of the Autonomous Treatment System Based on Machine Learning in patients with Covid-19, Post-Acute Sequelae of SARS-CoV-2 infection and influenza.

DETAILED DESCRIPTION:
This study has enrolled 27 patients diagnosed with Covid-19, Post-Acute Sequelae of SARS-CoV-2 infection, and influenza. Of these patients, 26 are outpatients, and 1 is hospitalized. After screening based on the inclusion and exclusion criteria, eligible patients will receive prescriptions recommended by the Autonomous Treatment System Based on Machine Learning in this observational trial.

The objectives of this study are:

1. To compare the classifications made by our machine learning system with those by physicians to assess the model's reliability and accuracy;
2. To evaluate Covid-19-related hospitalizations or deaths from any cause through day 28;
3. To determine if the machine learning system's recommended prescription alleviates symptoms of Covid-19, Post-Acute Sequelae of SARS-CoV-2 infection, and influenza;
4. To monitor participants who tested positive for the Covid-19 for 28 days after initiating treatment, looking for potential rebound cases.

Participants will use an online application to receive the recommended prescription results and will forward these results to a physician for verification. Patients are instructed to complete the online analysis every 3 days or whenever their symptoms change, whichever comes first. They are also asked to adhere to the prescribed medication regimen. Research physicians will conduct follow-ups with patients every 3 days via phone calls. The potential treatments patients may receive include any of the following Traditional Chinese Medicine formulas: LizCovidCure-1, LizCovidCure-2, LizCovidCure-3, LizCovidCure-4, and LizCovid-5.

ELIGIBILITY:
Inclusion Criteria:

* Either male or female (14 years or older), and their COVID-19 vaccination status was not a factor for inclusion.
* Subjects with any high-risk conditions
* Subjects with positive sars-cov-2 rapid antigen results in 30 days
* Subjects with post Covid-19 syndrome

Exclusion Criteria:

* pregnant individuals
* subjects with known histories of allergic reactions to medical herbs commonly used in Traditional Chinese Medicine (TCMs)

Ages: 14 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with active SARS-Cov-2 infection within 30 days patients with Post-Acute Sequelae of SARS-CoV-2 infection and patients with influenza.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Classification Accuracy | 1 Day
  compare the classifications made by our machine learning system with those by physicians, to assess the model's reliability

SECONDARY OUTCOMES:
Hospitalization Rate and Death | 28 Days
  we assess Covid-19-related hospitalization or death from any cause through day 28

OTHER OUTCOMES:
Symptom Alleviation | 28 Days
  Days of symptom disappearance
Re-infection Cases | 28 days
  Number of cases with recurrence-infection after treatment

CONTACTS AND LOCATIONS:
Overall Officials: jiale xian, MHA, Study Chair — Lizora LLC
Locations (1):
- Sheng'Ai Traditional Medicine Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
No plan to share the individual participant data (IPD).